CLINICAL TRIAL: NCT05027308
Title: A Phase 3, Open-label Safety Study of Teduglutide in Japanese Pediatric Patients With Short Bowel Syndrome Who Are Dependent on Parenteral Support, Aged 4 Months of Corrected Gestational Age or Older, and Requiring the Dosing of 1.25 mg Formulation
Brief Title: A Study of Teduglutide in Japanese Children With Short Bowel Syndrome Aged 4 Months or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-633-3008; U1111-1267-3327 (Other: WHO); jRCT2021210035 (Registry Identifier: jRCT); 2022-003572-16 (EudraCT Number)
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Short Bowel Syndrome
Keywords: Drug Therapy
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Teduglutide 0.05 milligram per kilogram (mg/kg) (Experimental): Participants will receive teduglutide 0.05 milligram per kilogram [mg/kg] (0.025 mg/kg for participants with moderate or greater renal impairment) subcutaneous [SC] injection once daily in a 28-week treatment cycle consisting of a 24-week treatment period followed by a 4-week no treatment follow-up period for a maximum of 3 cycles.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Teduglutide 0.05 mg/kg SC injection
  Other Names: TAK-633

SUMMARY:
The main aims of the study are to check for side effects from teduglutide.

Participants will receive a daily injection of teduglutide just under the skin (subcutaneous) for 24 weeks. Then they are followed up for another 4 weeks. Participants may be able to repeat this treatment if they meet specific criteria. The study doctors will check for side effects from teduglutide until it becomes commercially available. The maximum duration of treatment is approximately 51.3 weeks.

DETAILED DESCRIPTION:
A study of teduglutide in Japanese children with short bowel syndrome aged 4 months or older.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female pediatric patient of corrected gestational age 4 months or older.
2. Body weight at the time of screening and baseline visits of at least 5 kg and <10 kg for participants with normal renal function or mild renal impairment (estimated glomerular filtration rate >=50 mL/min/1.73 m^2), OR at least 10 kg and <20 kg for participants with moderate or greater renal impairment (estimated glomerular filtration rate <50 mL/min/1.73 m^2).
3. Diagnosis of short bowel syndrome (SBS) with intestinal failure, defined as dependence on PS to provide at least 30% of fluid or caloric needs.
4. Participants to have stable PS for at least 1 month prior to screening as assessed by the investigator. Stable PS is defined as inability to significantly reduce parenteral nutrition/intravenous fluid (PN/IV) support, usually associated with minimal or no advance in enteral feeds (ie, 10% or less change in PN or advance in feeds), assessed by the investigator.

Exclusion Criteria:

1. A parent/guardian who is not capable of understanding or not willing to adhere to the study visit schedule and other protocol requirements.
2. Clinically significant intestinal obstruction, active or recurrent pancreatic or biliary disease, or dysmotility that prevents the advancement of enteral intake.
3. Intestinal malabsorption due to a genetic condition, such as cystic fibrosis, microvillus inclusion disease, etc.
4. Severe, known dysmotility syndrome, such as pseudo-obstruction or persistent, severe, active gastroschisis-related dysmotility, that is the primary contributing factor to feeding intolerance and inability to reduce PS, prior to screening. Dysmotility is defined as severe if it is expected to limit the advancement of enteral feeding.
5. Major gastrointestinal (GI) surgical intervention including significant intestinal resection or bowel lengthening procedure within 3 months prior to screening (insertion of feeding tube, anastomotic ulcer repair, minor intestinal resections =<10 cm and endoscopic procedures are allowed).
6. Cardiac disease that makes the patient vulnerable to changes in fluid status.
7. History of cancer or known cancer predisposition syndrome, such as juvenile polyposis or Beckwith-Wiedemann syndrome, or first degree relative with early onset of GI cancer (including hepatobiliary and pancreatic cancer).
8. Concurrent treatment with glucagon-like peptide-2 (GLP-2), human growth hormone, or analogs of these hormones within 6 months prior to the screening visit, or concurrent treatment with octreotide, or GLP-1 analogs within 30 days prior to the screening visit.
9. Concurrent treatment with biological therapy (eg, anti-tumor necrosis factor [anti-TNF]) for active Crohn's disease within 6 months prior to the screening visit.
10. Participation in a clinical study using an experimental drug (other than glutamine or omegaven) within 3 months or 5.5 half-lives of the experimental drug, whichever is longer, prior to the screening visit and for the duration of the study.
11. Known or suspected intolerance or hypersensitivity to the study drug, closely related compounds, or any of the stated ingredients.
12. Signs of active, severe, or unstable clinically significant hepatic impairment during the screening period as meeting at least 2 of any of the following parameters:

    1. International normalized ratio >1.5 not corrected with parenteral vitamin K
    2. Platelet count <100×10^3/mcrL due to portal hypertension
    3. Presence of clinically significant gastric or esophageal varices
    4. Cirrhosis
    5. Persistent cholestasis defined as conjugated bilirubin >4 mg/dL (>68 mcr mol/L) over a 2-week period during screening
    6. Total bilirubin >=2x upper limit of normal (ULN)
    7. Aspartate aminotransferase (AST) >=3x ULN
    8. Alanine aminotransferase (ALT) >=3x ULN

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (6):
- Japan (6):
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Tohoku University Hospital, Sendai, Miyagi
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Akita University Hospital, Akita
  - Kyushu University Hospital, Fukuoka
  - Kagoshiha University Hospital, Kagoshima

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites).

REFERENCES:
- [Derived] Masumoto K, Muto M, Sasaki T, Shikamura M, Tanaka T, Sakui S, Miyamoto M, Nakano H, Kondo T, Ieiri S. Teduglutide in pediatric patients under 10 kg with short bowel syndrome on parenteral support: An open-label study. Pediatr Int. 2026 Jan-Dec;68(1):e70301. doi: 10.1111/ped.70301. PMID 41454663
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/613b9c47c61629002b6311f0

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants took part in the study at six investigative sites in Japan from 4 January 2022 to 27 September 2023.
Pre-assignment Details: Pediatric participants with a diagnosis of short bowel syndrome (SBS) dependent on parenteral support (PS) were enrolled in the study based on the eligibility criteria to receive teduglutide.
Groups:
- Teduglutide: Participants received teduglutide 0.05 milligram per kilogram [mg/kg] (0.025 mg/kg for participants with moderate or greater renal impairment) subcutaneous [SC] injection once daily in a 28-week treatment cycle consisting of a 24-week treatment period followed by a 4-week no treatment follow-up period for a maximum of 3 cycles.
Period: Overall Study
Arm/Group | Teduglutide
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3
Height for Age Z-Score at Baseline [Mean (Standard Deviation); unit: Z score] — A Z-score is the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). According to the World Health Organization (WHO) Child Growth Standards used for assessment of this characteristic, a height for age Z-score below -2 indicates stunted.
  Z score | -3.060 (1.1601)
Weight for Age Z-Score at Baseline [Mean (Standard Deviation); unit: Z score] — A Z-score is the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). According to WHO Child Growth Standards used for assessment of this characteristic, a weight for age Z-score below -2 indicates underweight.
  Z score | -3.017 (1.8048)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAEs were defined as any AEs whose onset occurred, severity worsened, or intensity increased after receiving the investigational product.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after end of treatment [EOT]/end of termination [ET] {up to 47.3-51.3 weeks})
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly /birth defect, is the other important medical event.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 3

3. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AESI, whether serious or non-serious, is one of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor may be appropriate.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs Reported as an Adverse Event
Description: Vital signs include systolic and diastolic blood pressure, heart rate and body temperature.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 0

5. Primary Outcome: Change From Baseline in Body Weight Z-Score at EOT
Description: A Z-score is the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). According to WHO Child Growth Standards used for assessment of this outcome measure, a weight for age Z-score below -2 indicates underweight.
Time Frame: Baseline, EOT (up to 47.3-51.3 weeks)
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Z score | 1.637 (2.8839)

6. Primary Outcome: Change From Baseline in Height Z-Score at EOT
Description: A Z-score is the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). According to WHO Child Growth Standards used for assessment of this outcome measure, a height for age Z-score below -2 indicates stunted.
Time Frame: Baseline, EOT (up to 47.3-51.3 weeks)
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Z score | 0.590 (1.9949)

7. Primary Outcome: Change From Baseline in Head Circumference Z-Score at EOT
Description: A Z-score is the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). According to the Food and Nutrition Technical Assistance (FANTA) Guide to Anthropometry used for assessment of this outcome measure, a head circumference for age Z-score below -2 indicates small head circumference.
Time Frame: Baseline, EOT (up to 47.3-51.3 weeks)
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Teduglutide
Number analyzed (Participants) | 2
Z score | 1.130 (0.4101)

8. Primary Outcome: Change From Baseline in Weight-for-Length Z-Score at EOT
Description: A Z-score is the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). According to WHO Child Growth Standards used for assessment of this outcome measure, a weight for length Z-score below -2 indicates wasted (recent and severe weight loss).
Time Frame: Baseline, EOT (up to 47.3-51.3 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Teduglutide
Number analyzed (Participants) | 1
Z score | 4.240 (NA) — The standard deviation was not estimable for a single participant.

9. Primary Outcome: Number of Participants With Any Laboratory Safety Finding Reported as an Adverse Event
Description: Laboratory safety parameters included biochemistry, hematology, and urinalysis.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 1

10. Primary Outcome: Number of Participants With a Change in Urine Output Reported as an Adverse Event
Description: Urine and stool output was recorded and calculated in the output diary over a 48-hour period of parenteral support (PS) and enteral nutrition (EN) stability before every site visit and within 1 week of implementing a change in the PS prescription.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 1

11. Primary Outcome: Number of Participants With a Change in Stool Output Reported as an Adverse Event
Description: Urine and stool output was recorded and calculated in the output diary over a 48-hour period of PS and EN stability before every site visit and within 1 week of implementing a change in the PS prescription.
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Population: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants | 0

12. Secondary Outcome: Change From Baseline in PS Volume
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume and calories during the treatment period. An end of treatment (EOT) was defined as the last determination of endpoint of the last cycle.
Time Frame: Baseline, Cycle 1 = Week 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 2: Week 0, 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 3 = Week 0, 1, 2, and EOT and overall EOT (for up to 47.3-51.3 weeks) [cycle length=28 weeks]
Population: Full Analysis Set included all enrolled participants, who were not screen failures, regardless of whether participants took any dose of teduglutide in the study. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: milliliters per kilograms (mL/kg)/day
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
milliliters per kilograms (mL/kg)/day
  Cycle 1, Week 1 | 3.13 (10.041)
  Cycle 1, Week 2 | 7.82 (19.334)
  Cycle 1, Week 4 | -1.31 (6.491)
  Cycle 1, Week 8 | 10.27 (13.788)
  Cycle 1, Week 12 | 5.83 (15.979)
  Cycle 1, Week 16 | 1.89 (16.386)
  Cycle 1, Week 20 | 1.82 (6.673)
  Cycle 1, Week 24 | 0.66 (9.511)
  Cycle 1, EOT | 0.66 (9.511)
  Cycle 2, Week 0 | -0.07 (12.808)
  Cycle 2 Week 1 | 0.11 (15.080)
  Cycle 2, Week 2 | -2.32 (13.465)
  Cycle 2, Week 4 | -0.71 (12.202)
  Cycle 2, Week 8 | -4.81 (13.214)
  Cycle 2, Week 12 | -8.42 (11.909)
  Cycle 2, Week 16 | -10.14 (10.452)
  Cycle 2, Week 20 | -8.20 (0.509)
  Cycle 2, Week 24: number analyzed (Participants) | 2
  Cycle 2, Week 24 | -9.28 (2.092)
  Cycle 2, EOT | -9.11 (1.508)
  Cycle 3, Week 0: number analyzed (Participants) | 1
  Cycle 3, Week 0 | -12.86 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, Week 1: number analyzed (Participants) | 1
  Cycle 3, Week 1 | -13.67 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, Week 2: number analyzed (Participants) | 1
  Cycle 3, Week 2 | -5.04 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, EOT: number analyzed (Participants) | 1
  Cycle 3, EOT | -5.04 (NA) — The standard deviation was not estimable for a single participant.
  Overall EOT | -10.99 (27.093)

13. Secondary Outcome: Percent Change From Baseline in PS Volume
Description: Percent change from baseline in PS volume was calculated as follows; (PS volume at each point [Week 1, 2, 4, 8, 12, 16, 20, 24, and EOT] - PS volume at baseline)/ PS volume at baseline *100 (percent). PS (parenteral nutrition or intravenous fluids) was to be considered for managing nutritional support in terms of volume and calories during the treatment period. An EOT was defined as the last determination of endpoint of the last cycle.
Time Frame: Baseline, Cycle 1 = Week 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 2 = Week 0, 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 3 = Week 0, 1, 2, and EOT and overall EOT (for up to 47.3-51.3 weeks) [cycle length=28 weeks]
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
percent change
  Cycle 1, Week 1 | 4.82 (13.391)
  Cycle 1, Week 2 | 11.27 (26.175)
  Cycle 1, Week 4 | -1.51 (8.881)
  Cycle 1, Week 8 | 13.48 (19.471)
  Cycle 1, Week 12 | 6.97 (22.006)
  Cycle 1, Week 16 | 1.61 (22.136)
  Cycle 1, Week 20 | 2.94 (8.794)
  Cycle 1, Week 24 | 1.24 (12.938)
  Cycle 1, EOT | 1.24 (12.938)
  Cycle 2, Week 0 | 0.07 (17.520)
  Cycle 2, Week 1 | 0.26 (20.634)
  Cycle 2, Week 2 | -2.81 (18.432)
  Cycle 2, Week 4 | -0.62 (16.671)
  Cycle 2, Week 8 | -6.00 (18.175)
  Cycle 2, Week 12 | -10.21 (16.645)
  Cycle 2, Week 16 | -13.03 (14.937)
  Cycle 2, Week 20 | -9.73 (3.073)
  Cycle 2, Week 24: number analyzed (Participants) | 2
  Cycle 2, Week 24 | -10.50 (6.059)
  Cycle 2, EOT | -10.98 (4.363)
  Cycle 3, Week 0: number analyzed (Participants) | 1
  Cycle 3, Week 0 | -17.69 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, Week 1: number analyzed (Participants) | 1
  Cycle 3, Week 1 | -18.79 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, Week 2: number analyzed (Participants) | 1
  Cycle 3, Week 2 | -6.93 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, EOT: number analyzed (Participants) | 1
  Cycle 3, EOT | -6.93 (NA) — The standard deviation was not estimable for a single participant.
  Overall EOT | -13.13 (37.259)

14. Secondary Outcome: Number of Participants Who Demonstrate at Least 20 Percent (%) Reduction From Baseline in PS Volume
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume and calories during the treatment period. An EOT was defined as the last determination of endpoint of the last cycle.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants
  Cycle 1, Week 1 | 0
  Cycle 1, Week 2 | 0
  Cycle 1, Week 4 | 0
  Cycle 1, Week 8 | 0
  Cycle 1, Week 12 | 0
  Cycle 1, Week 16 | 1
  Cycle 1, Week 20 | 0
  Cycle 1, Week 24 | 0
  Cycle 1, EOT | 0
  Cycle 2, Week 0 | 0
  Cycle 2, Week 1 | 1
  Cycle 2, Week 2 | 1
  Cycle 2, Week 4 | 0
  Cycle 2, Week 8 | 1
  Cycle 2, Week 12 | 1
  Cycle 2, Week 16 | 1
  Cycle 2, Week 20 | 0
  Cycle 2, Week 24: number analyzed (Participants) | 2
  Cycle 2, Week 24 | 0
  Cycle 2, EOT | 0
  Cycle 3, Week 0: number analyzed (Participants) | 1
  Cycle 3, Week 0 | 0
  Cycle 3, Week 1: number analyzed (Participants) | 1
  Cycle 3, Week 1 | 0
  Cycle 3, Week 2: number analyzed (Participants) | 1
  Cycle 3, Week 2 | 0
  Cycle 3, EOT: number analyzed (Participants) | 1
  Cycle 3, EOT | 0
  Overall EOT | 1

15. Secondary Outcome: Number of Participants Who Achieved Enteral Autonomy
Description: Achieving enteral autonomy is defined as complete weaning off PS. PS (parenteral nutrition or intravenous fluids) was to be considered for managing nutritional support in terms of volume and calories during the treatment period.
Time Frame: Cycle 1 = Week 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 2 = Week 0, 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 3 = Week 0, 1, 2, and EOT and overall EOT (for up to 47.3-51.3 weeks) [cycle length=28 weeks]
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
Participants
  Cycle 1, Week 1 | 0
  Cycle 1, Week 2 | 0
  Cycle 1, Week 4 | 0
  Cycle 1, Week 8 | 0
  Cycle 1, Week 12 | 0
  Cycle 1, Week 16 | 0
  Cycle 1, Week 20 | 0
  Cycle 1, Week 24 | 0
  Cycle 1, EOT | 0
  Cycle 2, Week 0 | 0
  Cycle 2, Week 1 | 0
  Cycle 2, Week 2 | 0
  Cycle 2, Week 4 | 0
  Cycle 2, Week 8 | 0
  Cycle 2, Week 12 | 0
  Cycle 2, Week 16 | 0
  Cycle 2, Week 20 | 0
  Cycle 2, Week 24: number analyzed (Participants) | 2
  Cycle 2, Week 24 | 0
  Cycle 2, EOT | 0
  Cycle 3, Week 0: number analyzed (Participants) | 1
  Cycle 3, Week 0 | 0
  Cycle 3, Week 1: number analyzed (Participants) | 1
  Cycle 3, Week 1 | 0
  Cycle 3, Week 2: number analyzed (Participants) | 1
  Cycle 3, Week 2 | 0
  Cycle 3, EOT: number analyzed (Participants) | 1
  Cycle 3, EOT | 0
  Overall EOT | 0

16. Secondary Outcome: Change From Baseline in Number of Days Per Week of PS Usage at EOT
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume and calories during the treatment period.
Time Frame: Baseline, Cycle 1 = Week 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 2 = Week 0, 1, 2, 4, 8, 12, 16, 20, 24, and EOT, Cycle 3 = Week 0, 1, 2, and EOT, and overall EOT (for 47.3-51.3 weeks) [cycle length=28 weeks]
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Teduglutide
Number analyzed (Participants) | 3
days per week
  Cycle 1, Week 1 | 0.0 (0.00)
  Cycle 1, Week 2 | 0.0 (0.00)
  Cycle 1, Week 4 | 0.0 (0.00)
  Cycle 1, Week 8 | 0.0 (0.00)
  Cycle 1, Week 12 | 0.0 (0.00)
  Cycle 1, Week 16 | 0.0 (0.00)
  Cycle 1, Week 20 | 0.0 (0.00)
  Cycle 1, Week 24 | 0.0 (0.00)
  Cycle 1, EOT | 0.0 (0.00)
  Cycle 2, Week 0 | 0.0 (0.00)
  Cycle 2, Week 1 | 0.0 (0.00)
  Cycle 2, Week 2 | 0.0 (0.00)
  Cycle 2, Week 4 | 0.0 (0.00)
  Cycle 2, Week 8 | 0.0 (0.00)
  Cycle 2, Week 12 | 0.0 (0.00)
  Cycle 2, Week 16 | 0.0 (0.00)
  Cycle 2, Week 20 | 0.0 (0.00)
  Cycle 2, Week 24: number analyzed (Participants) | 2
  Cycle 2, Week 24 | 0.0 (0.00)
  Cycle 2, EOT | 0.0 (0.00)
  Cycle 3, Week 0: number analyzed (Participants) | 1
  Cycle 3, Week 0 | 0.0 (0.00)
  Cycle 3, Week 1: number analyzed (Participants) | 1
  Cycle 3, Week 1 | 0.0 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, Week 2: number analyzed (Participants) | 1
  Cycle 3, Week 2 | 0.0 (NA) — The standard deviation was not estimable for a single participant.
  Cycle 3, EOT: number analyzed (Participants) | 1
  Cycle 3, EOT | 0.0 (NA) — The standard deviation was not estimable for a single participant.
  Overall EOT | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until follow-up visit (4 weeks after EOT/ET [up to 47.3-51.3 weeks])
Description: Safety Analysis Set included all participants who received at least 1 dose of study teduglutide.
Arm/Group | Teduglutide
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teduglutide (N=3)
Bacteraemia (Infections and infestations) | 1
Catheter site pruritus (General disorders) | 1
Device breakage (Product Issues) | 1
Device related infection (Infections and infestations) | 2
Vascular device occlusion (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teduglutide (N=3)
Blood iron increased (Investigations) | 1
COVID-19 (Infections and infestations) | 2
Catheter site rash (General disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 2
Lactic acidosis (Metabolism and nutrition disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 2
Skin candida (Infections and infestations) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT05027308/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT05027308/SAP_001.pdf